CLINICAL TRIAL: NCT06109779
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Global Study of Rilvegostomig in Combination With Chemotherapy as Adjuvant Treatment After Resection of Biliary Tract Cancer With Curative Intent (ARTEMIDE-Biliary01)
Brief Title: Rilvegostomig + Chemotherapy as Adjuvant Therapy for Biliary Tract Cancer After Resection (ARTEMIDE-Biliary01)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7025C00001; 2023-506054-20-00 (Other: EU Clinical Trial Number)
Record Dates: First submitted 2023-10-26; First posted 2023-10-31 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Biliary Tract Cancer
Keywords: Adenocarcinoma of the biliary tract; Biliary tract Cancer; Gall bladder cancer; Intrahepatic Cholangiocarcinoma; Distal Cholangiocarcinoma; Perihilar Cholangiocarcinoma; Klatskin Tumors; Bile duct cancer; Immunotherapy; Cholangiocarcinoma; Rilvegostomig; S-1; Gemcitabine/cisplatin; Capecitabine
MeSH Terms: conditions — Biliary Tract Neoplasms; Gallbladder Neoplasms; Cholangiocarcinoma; Klatskin Tumor; Bile Duct Neoplasms | interventions — Capecitabine; Gemcitabine; Cisplatin; S 1 (combination); Tegafur

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Rilvegostomig IV infusion + Investigator choice of chemotherapy (Capecitabine or Gemcitabine/Cisplatin or S-1)
  Interventions: Drug: Rilvegostomig; Drug: Capecitabine; Drug: Gemcitabine/Cisplatin; Drug: S-1 [Tegafur/Oteracil/gimeracil]
- Arm B (Placebo Comparator): Placebo IV infusion + Investigator choice of chemotherapy (Capecitabine or Gemcitabine/Cisplatin or S-1)
  Interventions: Drug: Placebo; Drug: Capecitabine; Drug: Gemcitabine/Cisplatin; Drug: S-1 [Tegafur/Oteracil/gimeracil]

INTERVENTIONS:
Drug: Rilvegostomig — Rilvegostomig IV (intravenous) Q3W
  Arms: Arm A
Drug: Placebo — Placebo IV (intravenous) Q3W
  Arms: Arm B
Drug: Capecitabine — Capecitabine (Oral) 1250 mg/m2 BID (twice daily) for 2 weeks on/1 week off in 21-day cycles or per local practice
Drug: Gemcitabine/Cisplatin — Gemcitabine/Cisplatin IV (Intravenous) 1000 mg/m2 plus cisplatin 25 mg/m2 on Day 1 and Day 8 of each 21-day cycle
Drug: S-1 [Tegafur/Oteracil/gimeracil] — S-1 [Tegafur/Oteracil/gimeracil] (Oral) BSA (body surface area)-based (40, 50, or 60 mg) BID for 4 weeks on 2 weeks off in 42-day cycles

SUMMARY:
A global study to assess the efficacy and tolerability of rilvegostomig compared to placebo in combination with investigator's choice of chemotherapy in participants with BTC after surgical resection with curative intent.

DETAILED DESCRIPTION:
This is a Phase III, randomized, double-blind, placebo-controlled, multicenter, global study to assess the efficacy and tolerability of rilvegostomig compared to placebo in combination with investigator's choice of chemotherapy (capecitabine, S-1(tegafur/ gimeracil/ oteracil) or gemcitabine/cisplatin) as adjuvant treatment in participants with BTC after resection with curative intent. This study will be conducted in patients with BTC who are at risk of recurrence after resection with curative intent.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the biliary tract (intrahepatic or extrahepatic cholangiocarcinoma (CCA) or muscle invasive gallbladder cancer (GBC)) after macroscopically complete resection (R0 or R1)
* Provision of a tumor sample collected at surgical resection.
* Randomization within 12 weeks after resection with adequate healing and removal of drains.
* Confirmed to be disease-free by imaging within 28 days prior to randomization.
* Eastern Cooperative Oncology Group performance status of 0 or 1

Exclusion Criteria:

* Participants with locally-advanced, unresectable, or metastatic disease at initial diagnosis.
* Ampullary cancer, neuroendocrine, mixed neuroendocrine and non-neuroendocrine neoplasms and nonepithelial tumors.
* Any anti-cancer therapy for BTC prior to surgery
* Active or prior documented autoimmune or inflammatory disorders or any severe or uncontrolled systemic disease
* Current or prior use of immunosuppressive medication within 14 days before the first dose
* Thromboembolic event within 3 months
* Active HBV or HCV infection unless treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2023-12-04 (Actual); Primary Completion 2029-01-02 (Estimated); Study Completion 2030-05-03 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival (RFS) for Arm A vs. Arm B | Approximately 5 years
  Recurrence-free survival (RFS) is defined as the time from randomization until the date of radiological recurrence guided by RECIST 1.1 or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) for Arm A vs. Arm B | up to 7 years
  Overall survival is defined as the time from randomization until the date of death due to any cause.

OTHER OUTCOMES:
Patient-reported tolerability Arm A vs. Arm B. | Up to approximately 7 years.
  Patient-reported tolerability is a multi-component endpoint defined as the proportion of participants in each arm reporting side effect bother, clinically meaningful impact on physical functioning and descriptive data on treatment-related symptoms.
Progression Free Survival (PFS) following recurrence Arm A vs. Arm B. | Up to approximately 7years
  Progression-free survival following recurrence is defined as the time from randomization until the earliest progression event after the start of the first subsequent therapy or death.

CONTACTS AND LOCATIONS:
Locations (176):
- United States (32):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, Newport Beach, California
  - Research Site, Orange, California
  - Research Site, Stanford, California
  - Research Site, West Hollywood, California
  - Research Site, Aurora, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Littleton, Colorado
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Altamonte Springs, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Iowa City, Iowa
  - Research Site, Kansas City, Kansas
  - Research Site, Lexington, Kentucky
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Grand Rapids, Michigan
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Commack, New York
  - Research Site, Mineola, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Dallas, Texas
  - Research Site, Tyler, Texas
  - Research Site, Vancouver, Washington
- Australia (5):
  - Research Site, Camperdown
  - Research Site, Clayton
  - Research Site, Murdoch
  - Research Site, Reservoir
  - Research Site, Westmead
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Edegem
  - Research Site, Leuven
- Brazil (6):
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Santa Maria
  - Research Site, Santo André
  - Research Site, São Paulo
  - Research Site, Vitória
- Canada (11):
  - Research Site, Vancouver, British Columbia
  - Research Site, Moncton, New Brunswick
  - Research Site, Halifax, Nova Scotia
  - Research Site, Brampton, Ontario
  - Research Site, Kingston, Ontario
  - Research Site, London, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
- China (24):
  - Research Site, Beijing
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Deyang
  - Research Site, Fuzhou
  - Research Site, Guangzhou
  - Research Site, Guiyang
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Hefei
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Lishui
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Nanning
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Zhengzhou
- Research Site, Herlev, Denmark
- France (8):
  - Research Site, Marseille
  - Research Site, Montpellier
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Rennes
  - Research Site, Strasbourg
  - Research Site, Toulouse
  - Research Site, Villejuif
- Germany (18):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Dortmund
  - Research Site, Dresden
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Esslingen A. N.
  - Research Site, Frankfurt
  - Research Site, Hamburg
  - Research Site, Heidelberg
  - Research Site, Leipzig
  - Research Site, Lübeck
  - Research Site, München
  - Research Site, Münster
  - Research Site, Stuttgart
  - Research Site, Tübingen
  - Research Site, Ulm
- Hong Kong (2):
  - Research Site, Hong Kong
  - Research Site, Shatin
- India (7):
  - Research Site, Delhi
  - Research Site, Kolkata
  - Research Site, Mumbai
  - Research Site, Mysuru
  - Research Site, New Delhi
  - Research Site, Vadodara
  - Research Site, Varanasi
- Italy (6):
  - Research Site, Florence
  - Research Site, Milan
  - Research Site, Padua
  - Research Site, Pisa
  - Research Site, Rozzano
  - Research Site, Tricase, Lecce
- Japan (14):
  - Research Site, Chūōku
  - Research Site, Hiroshima
  - Research Site, Kashiwa
  - Research Site, Kitaadachi-gun
  - Research Site, Kōtoku
  - Research Site, Mitaka-shi
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sendai
  - Research Site, Suita-shi
  - Research Site, Toyama
  - Research Site, Ube
  - Research Site, Wakayama
  - Research Site, Yokohama
- Research Site, Oslo, Norway
- Poland (8):
  - Research Site, Bydgoszcz
  - Research Site, Katowice
  - Research Site, Koszalin
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Przemyśl
  - Research Site, Tomaszów Mazowiecki
  - Research Site, Warsaw
- South Korea (2):
  - Research Site, Seongnam-si
  - Research Site, Seoul
- Spain (6):
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat
  - Research Site, Madrid
  - Research Site, Málaga
  - Research Site, Pamplona
  - Research Site, Santander
- Taiwan (5):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (5):
  - Research Site, Hat Yai
  - Research Site, Khon Kaen
  - Research Site, Muang
  - Research Site, Naimuang
  - Research Site, Si Sa Ket
- Turkey (Türkiye) (6):
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Erzurum
  - Research Site, Fatih-Istanbul
  - Research Site, Istanbul
  - Research Site, Samsun
- United Kingdom (6):
  - Research Site, Cambridge
  - Research Site, Edgbaston
  - Research Site, Glasgow, Scotland
  - Research Site, London
  - Research Site, Manchester
  - Research Site, Sutton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
URL: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure